CLINICAL TRIAL: NCT06336031
Title: Impact of Blood Phobia on Fainting Susceptibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Dr. Victoria Claydon, Professor, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 30002163
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Syncope, Vasovagal; Blood, Injection, Injury Type Phobia
Keywords: tilt table
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Calcium Channels, R-Type

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Image and video data set shown with BII stimuli. (Experimental): Participants will undergo this test on two separate days. On each day, participants will be asked to watch a series of videos and images. For this arm of the study, participants will view the BII phobia-related stimuli.
  Interventions: Other: blood-injection-injury (BII) phobia stimuli
- Image and video data set shown with neutral stimuli. (Placebo Comparator): Participants will undergo this test on two separate days. On each day, participants will be asked to watch a series of videos and images. For this arm of the study, participants will view the neutral stimuli.
  Interventions: Other: neutral stimuli

INTERVENTIONS:
Other: blood-injection-injury (BII) phobia stimuli — 498 seconds of BII phobia-related images and videos will begin two-minutes prior to head-up tilt test, while in supine.
  Arms: Image and video data set shown with BII stimuli.
Other: neutral stimuli — 498 seconds of neutral images and videos will begin two-minutes prior to head-up tilt test, while in supine.
  Arms: Image and video data set shown with neutral stimuli.

SUMMARY:
The primary purpose of this study is to characterize cardiovascular autonomic function to emotional stimuli (blood-injection-injury phobia [needle phobia]) during an orthostatic (upright) challenge in individuals with and without known needle phobia. It is well established that emotional stress can produce hypotensive (low blood pressure) reactions. Interestingly, these hypotensive reactions to venipuncture (even with minimal blood drawn), insulin injections, finger sticks for blood sugar monitoring, dental care, and vaccinations can affect up to a quarter of adults and appear to be uniquely associated with blood-injection-injury phobia rather than other phobias. These hypotensive reactions can ultimately lead to a vasovagal syncope (fainting) response, and lead to increased avoidance of medical and dental procedures as a result of this phobia. Ultimately, this has severe implications on public health and places additional strain on the Canadian healthcare system. Currently, there is limited understanding surrounding the initiation of this response. Additionally, a comprehensive profile of cardiovascular autonomic function during exposure to provoking stimuli during orthostatic stress has not been captured in the literature. We will test individuals with and without blood-injection-injury phobia using our standard approach while exposing them to emotional stimuli.

DETAILED DESCRIPTION:
The purpose of this study is to characterize cardiovascular autonomic function to emotional stimuli (blood-injection-injury phobia [needle phobia]) during an orthostatic (upright) challenge in individuals with and without known needle phobia. It is well established that emotional stress can produce hypotensive (low blood pressure) reactions. Interestingly, these hypotensive reactions to venipuncture (even with minimal blood drawn), insulin injections, finger sticks for blood sugar monitoring, dental care, and vaccinations can affect up to a quarter of adults and appear to be uniquely associated with blood-injection-injury phobia rather than other phobias. These hypotensive reactions can ultimately lead to a vasovagal syncope (fainting) response, and lead to increased avoidance of medical and dental procedures as a result of this phobia. Ultimately, this has severe implications on public health and places additional strain on the Canadian healthcare system. Currently, there is limited understanding surrounding the initiation of this response. Additionally, a comprehensive profile of cardiovascular autonomic function during exposure to provoking stimuli during orthostatic stress has not been captured in the literature. We will test individuals with and without blood-injection-injury phobia using our standard approach while exposing them to emotional stimuli.

Volunteers (n=20) will be asked to undergo a "tilt test" to assess cardiovascular reflex control and orthostatic tolerance (measured as time to presyncope, or near fainting, in minutes). We and others have previously shown this technique to be reproducible, reliable, and to have high sensitivity and specificity for differentiating persons with differing orthostatic tolerance, or for examining the effects of interventions aimed at improving orthostatic tolerance.

Volunteers will undergo the test on two separate days. On one test day (the order of which will be randomized) the volunteer will be shown a series of photos and videos during the upright tilt portion of the test. One day the series of content will consist of blood-injection-injury phobia content and the other day will have neutral content. Cardiovascular measures will be monitored through the test. The study will be conducted in a randomised fashion.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* 18 to 50 years old
* those without a suspected BII fear and those with a suspected fear
* english speaking

Exclusion Criteria:

* diagnosis of any cardiovacular or neurological disorder
* menopausal
* taking medication for a cardiovascular condition
* if they are pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Orthostatic Tolerance | 0-50 minutes
  Time (in minutes) to reach presyncope

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Claydon, PhD, Principal Investigator — Professor, Biomedical Physiology and Kinesiology
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be presented in aggregate form and no identifiers will be included.

REFERENCES:
- [Background] Trost Z, Jones A, Guck A, Vervoort T, Kowalsky JM, France CR. Initial validation of a virtual blood draw exposure paradigm for fear of blood and needles. J Anxiety Disord. 2017 Oct;51:65-71. doi: 10.1016/j.janxdis.2017.03.002. Epub 2017 Mar 16. PMID 28780134
- [Background] Stinson FS, Dawson DA, Patricia Chou S, Smith S, Goldstein RB, June Ruan W, Grant BF. The epidemiology of DSM-IV specific phobia in the USA: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Psychol Med. 2007 Jul;37(7):1047-59. doi: 10.1017/S0033291707000086. Epub 2007 Mar 5. PMID 17335637
- [Background] France CR, France JL, Himawan LK, Stephens KY, Frame-Brown TA, Venable GA, Menitove JE. How afraid are you of having blood drawn from your arm? A simple fear question predicts vasovagal reactions without causing them among high school donors. Transfusion. 2013 Feb;53(2):315-21. doi: 10.1111/j.1537-2995.2012.03726.x. Epub 2012 Jun 7. PMID 22670781
- [Background] Y. M. A. Al Shamma, R. Hainsworth, in Cardiogenic Reflexes. (Eds: R. Hainsworth, P.N. McWilliam, D.S.A.. Mary), OUP, Oxford, 1987, p. 431_ _-432.
- [Background] Brown CM, Hainsworth R. Forearm vascular responses during orthostatic stress in control subjects and patients with posturally related syncope. Clin Auton Res. 2000 Apr;10(2):57-61. doi: 10.1007/BF02279892. PMID 10823336
- [Background] Bush VE, Wight VL, Brown CM, Hainsworth R. Vascular responses to orthostatic stress in patients with postural tachycardia syndrome (POTS), in patients with low orthostatic tolerance, and in asymptomatic controls. Clin Auton Res. 2000 Oct;10(5):279-84. doi: 10.1007/BF02281110. PMID 11198483
- [Background] Claydon VE, Hainsworth R. Salt supplementation improves orthostatic cerebral and peripheral vascular control in patients with syncope. Hypertension. 2004 Apr;43(4):809-13. doi: 10.1161/01.HYP.0000122269.05049.e7. Epub 2004 Feb 23. PMID 14981050
- [Background] Claydon VE, Hainsworth R. Cerebral autoregulation during orthostatic stress in healthy controls and in patients with posturally related syncope. Clin Auton Res. 2003 Oct;13(5):321-9. doi: 10.1007/s10286-003-0120-8. PMID 14564654
- [Background] el-Bedawi KM, Hainsworth R. Combined head-up tilt and lower body suction: a test of orthostatic tolerance. Clin Auton Res. 1994 Apr;4(1-2):41-7. doi: 10.1007/BF01828837. PMID 8054836
- [Background] Cooper VL, Hainsworth R. Carotid baroreceptor reflexes in humans during orthostatic stress. Exp Physiol. 2001 Sep;86(5):677-81. doi: 10.1113/eph8602213. PMID 11571497
- [Background] Cooper VL, Hainsworth R. Effects of dietary salt on orthostatic tolerance, blood pressure and baroreceptor sensitivity in patients with syncope. Clin Auton Res. 2002 Aug;12(4):236-41. doi: 10.1007/s10286-002-0018-x. PMID 12357276
- [Background] Claydon VE, Schroeder C, Norcliffe LJ, Jordan J, Hainsworth R. Water drinking improves orthostatic tolerance in patients with posturally related syncope. Clin Sci (Lond). 2006 Mar;110(3):343-52. doi: 10.1042/CS20050279. PMID 16321141
- [Background] Schroeder C, Bush VE, Norcliffe LJ, Luft FC, Tank J, Jordan J, Hainsworth R. Water drinking acutely improves orthostatic tolerance in healthy subjects. Circulation. 2002 Nov 26;106(22):2806-11. doi: 10.1161/01.cir.0000038921.64575.d0. PMID 12451007